CLINICAL TRIAL: NCT01533779
Title: Neutrophil Extracellular Traps (NETs) Formation Following Chemotherapy for Pediatric Hematological and Solid Tumors, and Its Relation to Other Neutrophil Functions and the Role of NETs in Antitumor Activity
Brief Title: Neutrophil Extracellular Traps (NETs) Formation Following Chemotherapy and Their Role in Antitumor Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Max Planck Institute for Infection Biology (Other); Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0592-11-TLV
Record Dates: First submitted 2012-02-12; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Pediatric Solid Malignancies; Pediatric Hematological Malignancies
Keywords: children; malignancy; neutrophil; neutrophil extracellular traps; superoxide production; hydrogen peroxide production; chemotaxis; myeloperoxidase; immunosurveillance; cancer cell lines
MeSH Terms: conditions — Neoplasms; Chemotaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Examine neutrophil extracellular traps (NETs) formation, in relation to other neutrophil functions like chemotaxis, superoxide production, hydrogen peroxide production, and the presence of myeloperoxidase, in pediatric patients undergoing chemotherpy for solid and hematological malignancies. This data could shed new light on the mechanism responsible for the increased susceptibility to infection among these patients and aid in improving their prophylactic antimicrobial treatment.

NETs formation against tumor cell lines and their ability to kill tumor cells will also be examined. The finding of NETs activity against tumor cells could have a major contribution to the investigators understanding of the function of the immune system against cancer.

DETAILED DESCRIPTION:
Neutrophil function, including NETs formation, chemotaxis, superoxide production, hydrogen peroxide production, and the presence of myeloperoxidase, will be examined in 50 pediatric patientsundergoing chemotherapy for solid and hematological malignancies. Children with the following malignancies will be examined: acute lymphoblastic leukemia,acute myelogenous leukemia,Hodgkin's lymphoma,non-Hodgkin's lymphoma, primary bone sarcoma,rhabdomyosarcoma,non-rhabdomyosarcoma,neuroblastoma,Wilms' tumor,hepatoblastoma or hepatocellular carcinoma,germ cell tumors, and hystiocytosis. Also those with brain tumors such as medulloblastom,low grade glioma,high grade glioma,ependymoma,and embryonal and pineal region tumors. Data gathered on the patients will include background data (age, gender, ethnicity) and background diseases, data on current illness (histologic type, grade, stage, response treatment,infectious episodes), and on the use of ranulocyte-colony stimulating factor (G-CSF).

The following time points will be examined:

1. At diagnosis, before initiation of chemotherapy.
2. immediately before the 2nd course.
3. After the middle course.
4. A month after the last course.
5. Three months after the last course.
6. In acute myelogenous leukemia and acute lymphoblastic leukemia,time points also include the middle of the maintenance course and 3 months after the end of maintenance.

An additional blood examination will be used to examine NETs formation against tumor cell lines and their ability to kill tumor cells.

ELIGIBILITY:
Inclusion Criteria:

Included in the study were patients with:

* Acute lymphoblastic leukemia or acute myelogenous leukemia.
* Hodgkin's lymphoma or non-Hodgkin's lymphoma.
* Primary bone sarcoma, rhabdomyosarcoma, non-rhabdomyosarcoma, neuroblastoma, Wilms' tumor, hepatoblastoma or hepatocellular carcinoma, hystiocytosis, and germ cell tumors.
* Medulloblastoma, low grade glioma, high grade glioma, ependymoma, and embryonal and pineal region tumors.

Exclusion Criteria:

* A severe background disease that may affect Neutrophil function (e.g., diabetes, lupus).

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All pediatric patients from birth to 21 years, male and female, undergoing chemotherapy treatment for solid and hematological malignancies.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sivan Achituv, MD, Principal Investigator — The department of pediatric hemato-oncology, Dana Childrens' Hospital, Tel-Aviv Sourasky Medical Center, Tel-Aviv, Israel
Locations (1):
- Department of pediatric hemato-oncology, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel